CLINICAL TRIAL: NCT04904315
Title: An Exploratory, Multicenter, Observational Study to Examine RNA Biomarkers of Psoriasis Subjects Through the Application of the Mindera Kit Part 2 (STAMP-2).
Brief Title: Subjects Through the Application of the Mindera Kit Part 2
Acronym: STAMP-2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mindera Health (Industry)
Responsible Party: Sponsor
Other Study IDs: MND-20-PsCl-02
Record Dates: First submitted 2021-05-19; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mindera Kit — The entire duration of the study, including the screening period, will be approximately 16 weeks. Mindera Kit will be applied with applicator and left on the skin for 5 minutes, and once removed, the investigational product (IP) will be placed in a buffer solution, sealed, labeled and sent to Mindera for processing.
  Other Names: MK Patch, Microdermal Patch

SUMMARY:
A 16 week study to examine if baseline or on-therapy transcriptomics can be used to help predict selection of medications and provide new therapeutic targets for drug development in psoriasis subjects.

ELIGIBILITY:
Inclusion Criteria

1. Subject must have the ability to understand and sign written informed consent.
2. Subject must be an adult male or female adult who is ≥ 18 years of age at the time of screening.
3. Subject must be diagnosed with psoriasis by either a dermatologist or a rheumatologist, with the affected area of ≥ 2 centimeters in diameter.
4. Subjects must be treated with anti-TNF-α (or biosimilar) therapy once enrolled in the study.A two-week period is required to washout of the previous biologic when switching therapies.

Exclusion Criteria

1. Subject is unable or unwilling to give written informed consent and/or to comply with study procedures.
2. Subject has had usage of topical psoriasis treatments on study lesion within 2 weeks prior to baseline studyvisit and unwilling to washout.
3. Subjects currently treated with Hydroxychloroquine (Plaquenil), unless otherwise approved by Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects who are 18 years of age or older with a diagnosis of psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Observation of on therapy transcriptomics to potentially aid in new therapeutic targets | 16 weeks
  To examine if baseline or on-therapy transcriptomics can be used to help predict selection of medications and provide new therapeutic targets for drug development in psoriasis subjects by collecting RNA and examining changes in PASI scores at the Week 4, 12, and 16 timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Toby Dickerson, Study Chair — CSO

IPD SHARING:
Plan to Share IPD: No
In order to protect patient privacy genetic data will not be shared outside of the study without further patient consent to do so. If other researchers would like access to the data they must reach out to the patients themselves.